CLINICAL TRIAL: NCT00685399
Title: An Open-label Proof-of-concept Study With a Double-masked, Dose-ranging Component to Assess the Effects of AIN457 in Patients With Noninfectious Uveitis
Brief Title: Safety and Efficacy of AIN457 in Noninfectious Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2208; 2011-001243-67 (EudraCT Number)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Non-infectious Uveitis
Keywords: Uveitis; eye; IL-17; IL-17A; IL17; AIN457; Vogt-Koyanagi-Harada; Behcet's; Behcet; Sympathetic ophthalmia; Multifocal choroiditis; Birdshot; HLA-B27; Birdshot retinochoroiditis; Retinal vasculitis; Sarcoidosis; Intermediate uveitis; Panuveitis; Posterior uveitis
MeSH Terms: conditions — Uveitis; Behcet Syndrome; Ophthalmia, Sympathetic; Multifocal Choroiditis; Birdshot Chorioretinopathy; Retinal Vasculitis; Sarcoidosis; Uveitis, Intermediate; Panuveitis; Uveitis, Posterior | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (Experimental): Participants were administered with AIN457 (Sp2/0derived) 10 milligrams per kilogram (mg/kg) intravenous (i.v.) dose on Day 1 and Day 22.
  Interventions: Drug: AIN457
- Cohort 2 (Experimental): Participants were administered with AIN457 (Sp2/0 or Chinese hamster ovary cell (CHO) derived) 10 mg/kg, (CHO derived) 3 mg/kg or (CHO derived) 1 mg/kg i.v. dose on Day 1 and if needed a second dose of AIN457 10 mg/kg i.v. dose either on Day 15 or Day 22. 3 participants from cohort 1 rolled on into this cohort.
  Interventions: Drug: AIN457
- Cohort 3 (Experimental): Participants were administered with AIN457 10 mg/kg i.v. dose on Day 1 and Day 22.
  Interventions: Drug: AIN 457
- Cohort 4 (Experimental): Extension period: Participants were administered with AIN457 10 mg/kg, i.v. (with or without a short course of corticosteroids) once a flare had occurred, or periodically at a frequency of not more than once per month at the discretion of the investigator.
  Interventions: Drug: AIN 457
- Cohort 5 (Experimental): Participants were administered with AIN457 30 mg/kg single i.v. dose. A second dose was given when all 4 participants completed at least 29 days, and the 30 mg/kg dose was well tolerated by all.
  Interventions: Drug: AIN457
- Cohort 6 Arm 1 (Experimental): Participants were administered with AIN457 300 mg subcutaneously (s.c.) and saline i.v. infusion every two weeks (Days 1, 15, 29, and 43).
  Interventions: Drug: AIN457
- Cohort 6 Arm 2 (Experimental): Participants were administered with AIN457 10 mg/kg i.v. and s.c. saline injections every two weeks (Days 1, 15, 29, and 43).
  Interventions: Drug: AIN 457
- Cohort 6 Arm 3 (Experimental): Participants were administered with AIN457 30 mg/kg i.v. and s.c. saline injections every 4 weeks (Days 1 and 29) and saline i.v. infusions and saline s.c. injections on Days 15 and 43 to maintain masking of treatment groups.
  Interventions: Drug: AIN457

INTERVENTIONS:
Drug: AIN457 — AIN457 subcutaneous dose
  Other Names: Secukinumab
  Arms: Cohort 1; Cohort 2
Drug: AIN 457 — AIN457 low dose (i.v)
  Other Names: Secukinumab
  Arms: Cohort 3; Cohort 4; Cohort 6 Arm 2
Drug: AIN457 — AIN457 high dose (i.v)
  Other Names: Secukinumab
  Arms: Cohort 5; Cohort 6 Arm 1; Cohort 6 Arm 3

SUMMARY:
This study was performed to evaluate the efficacy and safety of AIN457 for patients with active uveitis that requires systemic immunosuppression.

ELIGIBILITY:
Inclusion criteria:

* Active uveitis (i.e., uveitis that is not in remission).
* Intermediate uveitis, posterior uveitis, or panuveitis must be sufficiently severe that systemic immunosuppression is indicated.

Exclusion criteria:

* Active infection.
* Weight must not be greater that 120kg.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (19):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigative Site, Littleton, Colorado
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Slingerlands, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Houston, Texas
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Letko E, Yeh S, Foster CS, Pleyer U, Brigell M, Grosskreutz CL; AIN457A2208 Study Group. Efficacy and safety of intravenous secukinumab in noninfectious uveitis requiring steroid-sparing immunosuppressive therapy. Ophthalmology. 2015 May;122(5):939-48. doi: 10.1016/j.ophtha.2014.12.033. Epub 2015 Jan 29. PMID 25638011
- [Derived] Hueber W, Patel DD, Dryja T, Wright AM, Koroleva I, Bruin G, Antoni C, Draelos Z, Gold MH; Psoriasis Study Group; Durez P, Tak PP, Gomez-Reino JJ; Rheumatoid Arthritis Study Group; Foster CS, Kim RY, Samson CM, Falk NS, Chu DS, Callanan D, Nguyen QD; Uveitis Study Group; Rose K, Haider A, Di Padova F. Effects of AIN457, a fully human antibody to interleukin-17A, on psoriasis, rheumatoid arthritis, and uveitis. Sci Transl Med. 2010 Oct 6;2(52):52ra72. doi: 10.1126/scitranslmed.3001107. PMID 20926833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-center study which comprised of 6 cohorts. This study was a proof of concept study.
Groups:
- Cohort 1: Participants were administered with AIN457 (Sp2/0-derived) 10 milligrams per kilogram (mg/kg) intravenous (i.v.) dose on Day 1 and Day 22.
- Cohort 2: Participants were administered with AIN457 (Sp2/0 or Chinese hamster ovary cell (CHO) derived) 10 mg/kg, (CHO-derived) 3 mg/kg or (CHO derived) 1 mg/kg i.v. dose on Day 1 and if needed a second dose of AIN457 10 mg/kg i.v. dose either on Day 15 or Day 22. 3 participants from cohort 1 rolled on into this cohort.
- Cohort 4: Participants who experienced a remission of their uveitis within 8 weeks after receiving their final dose of AIN457 while enrolled in Cohorts 1, 2, 3, 5 or 6 were administered with AIN457 10 mg/kg, i.v. infusion (with or without a short course of corticosteroids) once a flare had occurred, or periodically at a frequency of not more than once per month at the discretion of the investigator.
Period: Treatment Period 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Started | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Started | 0 | 14 | 5 | 0 (in extension period only) | 4 | 12 | 13 | 12
Completed | 0 | 2 | 2 | 0 (in extension period only) | 4 | 10 | 13 | 10
Not Completed | 0 | 12 | 3 | 0 | 0 | 2 | 0 | 2
Not completed — Administrative Problems | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 10 | 2 | 0 | 0 | 1 | 0 | 0
Period: Extension
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Started | 0 | 0 | 0 | 28 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0
Not completed — Administrative Issues | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants were administered with AIN457 (Sp2/0-derived) 10 mg/kg i.v. dose on Day 1 and Day 22.
- Cohort 2: Participants were administered with AIN457 (Sp2/0 or CHO derived) 10 mg/kg, (CHO-derived) 3 mg/kg or (CHO derived) 1 mg/kg i.v. dose on Day 1 and if needed second dose of AIN457 10 mg/kg i.v. dose either on Day 15 or Day 22. 3 participants from cohort 1 rolled on into this cohort.
- Cohort 6 Arm 1: Participants were administered with AIN457 300 mg s.c. and saline i.v. infusion every two weeks (Days 1, 15, 29, and 43).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3 | Total
Number analyzed (Participants) | 16 | 14 | 5 | 4 | 12 | 13 | 12 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 15 | 13 | 5 | 4 | 12 | 11 | 12 | 72
  >=65 years | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 3 | 3 | 8 | 9 | 9 | 54
  Male | 4 | 4 | 2 | 1 | 4 | 4 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 0 | 0 | 2 | 2 | 3 | 13
  White | 7 | 10 | 4 | 1 | 9 | 9 | 8 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 1 | 2 | 1 | 2 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Who Died
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: Day 1 to Day 603
Population: Safety Analysis Set (SAS) consisted of all participants who received at least one dose of study drug and had at least one post-baseline safety assessment. All safety evaluations were carried out on the safety analysis set.
Measure: Number; unit: participants
Groups:
- Cohort 4: Participants were administered with AIN457 10 mg/kg, i.v. (with or without a short course of corticosteroids) once a flare had occurred, or periodically at a frequency of not more than once per month at the discretion of the investigator.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Number analyzed (Participants) | 16 | 17 | 5 | 28 | 4 | 12 | 13 | 12
participants
  SAEs | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs | 15 | 12 | 5 | 23 | 3 | 10 | 10 | 12

2. Secondary Outcome: Number of Responders in Cohort 1, 2, 3 and 6 at Day 57
Description: A "responder" was defined as a participant who fulfilled at least one of the 3 criteria compared to baseline: 1. Increase in visual acuity by at least 15 letters using Early Treatment Diabetic Retinopathy Study method, no increase in daily prednisone dose compared to week 1 and without worsening of uveitis. 2. Decrease in vitreous haze by 2 steps or more or for participants with anterior uveitis, resolution of the anterior chamber inflammation (i.e., no cells or only a rare cell in the anterior chamber (score 0 or trace (0.5+)), use measurement before dilation), no increase in daily prednisone dose compared to week 1 and without any worsening of uveitis.3 For those participant on a. >20 mg/day of prednisone during week 1: Reduction in daily prednisone dose to 10 mg/day or less. b. ≤20 mg/day of prednisone during week 1: Reduction in daily prednisone dose to 0 mg/day. c. topical corticosteroids during week 1: Reduction in daily topical corticosteroid dose to 0 during the last 2 weeks.
Time Frame: Day 1 (Baseline), Day 57
Population: The Per Protocol Analysis Set (PPAS) consisted of all participants who received study drug, completed the treatment phase of the trial without clinically significant protocol deviations and have at least one post-baseline assessment for one of the outcomes that define participants who respond.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Number analyzed (Participants) | 15 | 14 | 5 | 12 | 13 | 11
Participants
  Intermediate uveitis | 0 | 1 | 0 | 1 | 1 | 3
  Pars planitis | 0 | 0 | 0 | 0 | 0 | 0
  Posterior uveitis | 3 | 0 | 0 | 1 | 2 | 0
  Panuveitis | 5 | 4 | 0 | 2 | 5 | 5
  Anterior uveitis | 3 | 1 | 0 | 0 | 0 | 0
  Birdshot | 0 | 0 | 2 | 0 | 0 | 0
  Sympathetic ophthalmia | 0 | 0 | 1 | 0 | 0 | 0
  Multi-focal choroiditis | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Complete Responders in Cohort 2, 3 and 6 at Day 57
Description: A "complete responder" was defined as a participant who was able to stop all topical and systemic corticosteroids in both eyes and maintain remission of uveitis (=remains a responder as defined above) lasting at least 1 week (since stopping corticosteroids, if corticosteroids were given).
Time Frame: Day 1 (Baseline), Day 57
Population: PPAS consisted of all participants who received study drug, completed the treatment phase of the trial without clinically significant protocol deviations and have at least one post-baseline assessment for one of the outcomes that define participants who respond.
Measure: Number; unit: Participants
Arm/Group | Cohort 2 | Cohort 3 | Cohort 6 Arm 1 | Cohort 6 Arm 2 | Cohort 6 Arm 3
Number analyzed (Participants) | 14 | 5 | 12 | 13 | 11
Participants
  Intermediate uveitis | 0 | 0 | 0 | 1 | 1
  Panuveitis | 1 | 0 | 1 | 2 | 2
  Pars planitis | 0 | 0 | 0 | 0 | 0
  Anterior uveitis | 1 | 0 | 0 | 0 | 0
  Birdshot | 0 | 2 | 0 | 0 | 0
  Sympathetic ophthalmia | 0 | 1 | 0 | 0 | 0
  Multi-focal choroiditis | 0 | 0 | 0 | 0 | 0
  Posterior uveitis | 0 | 0 | 1 | 2 | 0

4. Secondary Outcome: Number of Participants With Reduction in Oral Prednisone or Topical Corticosteroid and Other Immunosuppressant Drugs
Description: Participants intake of oral prednisone or topical corticosteroid and other immunosuppressant drugs was reduced if participant was on up to 1.5 mg/kg/day dose of prednisone during the week prior to Day 1 or whom the resumption of prednisone was not considered the appropriate systemic therapy by investigator or who have never been on systemic immunosuppressive therapy and whose uveitis was so severe that, in the clinician's judgment, prednisone at a dose of 1.0-1.5 mg/kg/day alone will be insufficient to control the uveitis or participant with HLA-B27-associated anterior uveitis who would ordinarily be started on systemic prednisone. The analysis was not conducted due to small sample size, insufficient number of participants and low initial doses; limited conclusions were drawn about dose response relationship leading to non summarization of results.
Time Frame: Baseline (Day 1) up to Month 8
Population: as for outcome 3
Groups:
- Complete Study: All participants who received study drug, completed the treatment phase of the trial without clinically significant protocol deviations and have non-missing values at both Day 1 and Day 57 for at least one of the outcomes that define participants who respond.
Arm/Group | Complete Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Were Able to Induce a Remission in Uveitis
Description: Participants with uveitis who were able to stop all topical and systemic topical corticosteroids in both eyes by Day 57 visit after the first course of one or two doses of AIN457 were to be categorized as nonresponders and were to be discontinued from the study at the Day 85 visit. The analysis was not conducted due to small sample size, insufficient number of participants and low initial doses; limited conclusions were drawn about dose response relationship leading to non summarization of results.
Time Frame: Day 1 to Day 85
Population: as for outcome 3
Arm/Group | Complete Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Remission in Uveitis
Description: Participants with uveitis who were able to stop all topical and systemic topical corticosteroids in both eyes after the first course of one or two doses by Day 57 visit . The analysis was not conducted due to small sample size, insufficient number of participants and low initial doses; limited conclusions were drawn about dose response relationship leading to non summarization of results.
Time Frame: Baseline (Day 1) up to Month 8
Population: as for outcome 3
Arm/Group | Complete Study
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Were Able to Re-induce a Remission if a Flare-up Occurs
Description: A flare was defined as an increase of inflammation in either eye so that the anterior chamber cell score or the vitreous haze score become 1+ or greater. Vitreous haze was evaluated with an indirect ophthalmoscope and a hand-held 20-diopter lens. Haze is defined as a reduction in the clarity of fundus details seen through the vitreous, the degree of haze was quantified using standard National Eye Institute (NEI) photographs. The standard photographs provide a grading scale with photographs of fundi with vitreous haze grades "0" (zero), "trace" (which counts as 0.5+), 1+, 2+, 3+, and 4+. If the amount of vitreous haze appears to fall between two integer grades, the value would be recorded as halfway between the grades. The analysis was not conducted due to small sample size, insufficient number of participants and low initial doses; limited conclusions were drawn about dose response relationship leading to non summarization of results.
Time Frame: Day 1 to Day 57
Population: as for outcome 3
Arm/Group | Complete Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 603 (End of study)
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects.
Groups:
- Cohort 2: Participants were administered with AIN457 (Sp2/0 or CHO derived) 10 mg/kg, (CHO-derived) 3 mg/kg or (CHO derived) 1 mg/kg i.v. dose on Day 1 and if needed second dose of AIN457 10 mg/kg i.v. dose either on Day 15 or Day 22.
- Cohort 6 - Arm 1: Participants were administered with AIN457 300 mg s.c.and saline i.v. infusion every two weeks (Days 1, 15, 29, and 43).
- Cohort 6 - Arm 2: Participants were administered with AIN457 10 mg/kg i.v. and s.c. saline injections every two weeks (Days 1, 15, 29, and 43).
- Cohort 6 - Arm 3: Participants were administered with AIN457 30 mg/kg i.v. and s.c. saline injections every 4 weeks (Days 1 and 29) and saline i.v. infusions and saline s.c. injections on Days 15 and 43 to maintain masking of treatment groups.
- Cohort 4 (Extension): Participants were administered with AIN457 10 mg/kg, i.v. (with or without a short course of corticosteroids) once a flare had occurred, or periodically at a frequency of not more than once per month at the discretion of the investigator.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6 - Arm 1 | Cohort 6 - Arm 2 | Cohort 6 - Arm 3 | Cohort 4 (Extension)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/5 | 0/4 | 0/12 | 0/13 | 0/12 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 1/5 | 0/4 | 1/12 | 0/13 | 0/12 | 1/28
Other Adverse Events (participants affected / at risk) | 15/16 | 12/17 | 5/5 | 3/4 | 9/12 | 10/13 | 12/12 | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=16) | Cohort 2 (N=17) | Cohort 3 (N=5) | Cohort 5 (N=4) | Cohort 6 - Arm 1 (N=12) | Cohort 6 - Arm 2 (N=13) | Cohort 6 - Arm 3 (N=12) | Cohort 4 (Extension) (N=28)
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=16) | Cohort 2 (N=17) | Cohort 3 (N=5) | Cohort 5 (N=4) | Cohort 6 - Arm 1 (N=12) | Cohort 6 - Arm 2 (N=13) | Cohort 6 - Arm 3 (N=12) | Cohort 4 (Extension) (N=28)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anterior chamber flare (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colour blindness acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye pain (Eye disorders) | 3 | 2 | 1 | 0 | 1 | 1 | 1 | 3
Eye pruritus (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Iris adhesions (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iris bombe (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Macular oedema (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scleritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Vision blurred (Eye disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 3 | 1
Visual acuity reduced (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 4
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 3 | 6
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil percentage increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein urine (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 10 | 4 | 3 | 2 | 5 | 3 | 4 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.